CLINICAL TRIAL: NCT00534560
Title: Multi-Centre, Parallel Group, Double-Blind, Placebo Controlled, Dose Ranging Study of the Efficacy and Tolerability of Tonabersat in the Prophylaxis of Migraine Headache and Open Label Extension
Brief Title: Dose Ranging Study of the Efficacy and Tolerability of Tonabersat in the Prophylaxis of Migraine Headache
Acronym: TEMPUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minster Research Ltd (Industry)
Responsible Party: Development Director, Minster Research Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TON/03/07-CLIN
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Migraine Without Aura; Migraine With Aura
MeSH Terms: conditions — Migraine without Aura; Migraine with Aura | interventions — tonabersat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Tonabersat
- 2 (Experimental)
  Interventions: Drug: Tonabersat
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tonabersat — Tablets, 4 week dose titration and 16 weeks treatment at target dose of 40 mg per day
  Other Names: SB220453
  Arms: 1
Drug: Tonabersat — Tablets: 4 week titration and 16 weeks at target dose of 80 mg per day
  Other Names: SB220453
  Arms: 2
Drug: Placebo — Tablets; 4 week dose titration with 16 weeks at target dose
  Arms: 3

SUMMARY:
Primary objective:

To investigate the efficacy and tolerability of two doses of tonabersat compared to placebo in the prophylaxis of migraine headache and to evaluate the longer term tolerability of tonabersat in an open label extension.

Secondary objective(s):

To obtain further data on the efficacy and dose response of tonabersat; To extend the safety and tolerability database of tonabersat; To obtain data on the pharmacokinetics of tonabersat.

DETAILED DESCRIPTION:
A multi-centre, double-blind, placebo controlled, randomized, parallel group, dose ranging study to investigate the efficacy and tolerability of two different target doses of tonabersat and placebo in the prophylaxis of migraine. Following initial screening patients will enter a 4 week baseline assessment period, prior to randomization to one of three treatment groups. Subsequently patients will be allocated, according to the predetermined randomization schedule, to treatment with placebo or a target dose of tonabersat 40 mg/day or 80 mg/day in a 20 week treatment period. A dose titration regimen will be employed over a period of 4 weeks and treatment will then be maintained for a further 16 weeks. During the baseline assessment period and the treatment period patients will maintain a daily record (diary data) of the occurrence of migraine headache, the severity of an attack, the presence/absence of a preceding aura, other symptoms associated with the migraine and details of the use of rescue medication (patients will be permitted to use their usual symptomatic/acute treatment as rescue medication throughout the trial). Patients will attend the clinic for assessment and collection of blood and urine samples for laboratory analysis, and a sub-population of patients will participate in a pharmacokinetic study. A total of 7 visits are planned during the randomized double-blind treatment period.

On completion of the randomized double-blind treatment period all patients will be offered the opportunity to enter an open label extension study where all patients receive tonabersat. A dose titration regimen will be employed over a period of 1 month and the final assigned dose of tonabersat (40, 60 or 80 mg/day) will be continued for the next 12 months. During the open label extension patients will attend the clinic for regular assessment of migraine status and safety. A total of 5 visits are planned.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated written informed consent is obtained prior to participation.
* Male or female patients between 18-65 years of age who are ambulatory and able to travel to the clinic; women of childbearing potential must be using a reliable form of contraception (contraceptive pill or double-barrier contraception - partner using condom and patient using spermicide, diaphragm, intra-uterine device or contraceptive sponge) for at least 2 months prior to enrolment and have a negative pregnancy test at screening. Women of childbearing potential must continue to practice birth control during and for at least two months after the study
* Patients with an established history of migraine of at least 1 year with or without aura meeting the diagnostic criteria of the International Classification of Headache Disorders - Edition 2.
* Patients should have experienced an average of at least 4 migraine attacks per month over the 3 months prior to entering the trial and at least 3 migraine attacks during the baseline period. Patients should report a maximum of 12 migraine headache days during the baseline period.

Exclusion Criteria:

* Patients with an onset of migraine according to the above criteria at age 50 years or more.
* Patients who experience > 12 headache days during the baseline period.
* Patients who have failed to respond to adequate trials of 3 or more preventive medications.
* Overuse of acute migraine treatments defined as ≥ 15 medication days per month of which no more than 9 days includes ergots or triptans.
* Any woman who is pregnant, lactating or not using medically acceptable contraception.
* Patients taking other medications used as prophylaxis for migraine including topiramate, methysergide, anti-spasticity agents (e.g. tizanidine) and new generation antipsychotics (e.g. olanzapine) currently or within 1 month prior to entry to the trial.
* Patients taking any of the following medications: beta-blockers, tricyclic antidepressants, antiepileptic drugs, calcium channel blockers, or monoamine oxidase inhibitors during or within 1 month prior to the study; daily oral NSAIDs, daily paracetamol, high dose magnesium supplements (600 mg/day), daily multivitamin preparations containing more than 10 mg riboflavin, daily use of oral corticosteroids, herbal preparations (e.g. feverfew, butterwort and St John's Wort). Patients who have received parenteral administration of botulinum toxin within the previous 3 months will also be excluded.
* Patients who, in the opinion of the Investigator, have significant cerebrovascular disease (e.g. transient ischemic attacks, stroke) or significant cardiovascular disease within 30 days prior to screening.
* Patients suffering from any significant psychiatric disorder.
* Patient has a concomitant disease or condition that, in the opinion of the Investigator, could interfere with the conduct of the study or could put the patient at unacceptable risk.
* Patients with renal dysfunction, defined as a serum creatinine of greater then 2 mg/dL.
* Patients with hepatic dysfunction defined as a liver function test (AST, ALT, alkaline phosphatase, bilirubin) of greater than twice the upper limit of normal for their age group.
* Patients with known alcohol or other substance abuse.
* Patient is a participating Investigator, sub-investigator, study coordinator, or employee of a participating Investigator, or is an immediate family member of the aforementioned.
* Any factor, which in the opinion of the Investigator would jeopardize the evaluation or safety or be associated with poor adherence to the protocol.
* The patient's primary care physician recommends the patient should not take part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Reduction in the mean monthly number of migraine attacks over the last 2 months of the treatment period. | 4 weeks baseline and 20 weeks DB treatment
Safety and tolerability: incidence of all AEs, serious adverse events (SAEs) and those leading to withdrawal of study medication, review of laboratory data, including hematology, biochemistry, and urinalysis, physical examinations, and vital signs. | 4 weeks baseline, 20 weeks DB treatment and 13 months open label extension
Assessment of population pharmacokinetics for tonabersat - blood samples will be collected from a sub-population of patients | 20 weeks DB treatment

SECONDARY OUTCOMES:
• Reduction in mean monthly migraine attacks during the last 4 months of the treatment period and during each month of the treatment period. | 4 weeks baseline and 20 weeks DB treatment
• Proportion of patients defined as a responder i.e. difference between treatment groups in the number of patients with a reduction of at least 50% in the mean monthly frequency of migraine attacks during defined periods. | 4 week baseline and 20 weeks DB treatment
• Reduction in mean monthly migraine headache days i.e. the difference between the two treatment groups in the reduction from baseline during defined periods | 4 weeks baseline and 20 weeks DB treatment
• Proportion of patients defined as a responder i.e. difference between treatment groups in the number of patients with a reduction of at least 50% in the mean monthly number of migraine headache days during defined periods | 4 weeks baseline and 20 weeks DB treatment
• Reduction in mean monthly consumption (number of days per month) of rescue medication during defined periods | 4 weeks baseline and 20 weeks DB treatment
• Onset of action (defined as first monthly period for which a significant difference between treatment groups is observed and is then maintained over the rest of the treatment period). | 4 weeks baseline and 20 weeks DB treatment
• Difference between treatment groups in the maximum severity of migraine attacks occurring during defined periods | 4 weeks baseline and 20 weeks DB treatment
• Summary of the Migraine Disability Assessment Score (MIDAS) assessments. | 4 weeks baseline, 20 weeks DB treatment and 13 months open label extension

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lipton, MD, Principal Investigator — Montefiore Medical Center Headache Unit

REFERENCES:
- [Background] Tfelt-Hansen P, Block G, Dahlof C, Diener HC, Ferrari MD, Goadsby PJ, Guidetti V, Jones B, Lipton RB, Massiou H, Meinert C, Sandrini G, Steiner T, Winter PB; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: second edition. Cephalalgia. 2000 Nov;20(9):765-86. doi: 10.1046/j.1468-2982.2000.00117.x. No abstract available. PMID 11167908
- [Background] Grosser K, Oelkers R, Hummel T, Geisslinger G, Brune K, Kobal G, Lotsch J. Olfactory and trigeminal event-related potentials in migraine. Cephalalgia. 2000 Sep;20(7):621-31. doi: 10.1111/j.1468-2982.2000.00094.x. PMID 11128819
- [Background] Hu XH, Markson LE, Lipton RB, Stewart WF, Berger ML. Burden of migraine in the United States: disability and economic costs. Arch Intern Med. 1999 Apr 26;159(8):813-8. doi: 10.1001/archinte.159.8.813. PMID 10219926
- [Background] Stewart WF, Lipton RB, Whyte J, Dowson A, Kolodner K, Liberman JN, Sawyer J. An international study to assess reliability of the Migraine Disability Assessment (MIDAS) score. Neurology. 1999 Sep 22;53(5):988-94. doi: 10.1212/wnl.53.5.988. PMID 10496257